CLINICAL TRIAL: NCT03674931
Title: Train the Brain With Music: Brain Plasticity and Cognitive Benefits Induced by Musical Practice in Elderly People in Germany and Switzerland
Brief Title: Train the Brain With Music: Brain Plasticity and Cognitive Benefits Induced by Musical Practice in Elderly People
Acronym: TBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Collaborators: Swiss National Science Foundation (Other); German Research Foundation (Other)
Responsible Party: Principal Investigator, Clara E James, Full Professor, School of Health Sciences Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81185
Record Dates: First submitted 2018-07-06; First posted 2018-09-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Age-related Cognitive Decline
Keywords: countervail age-related cognitive and cerebral decline; healthy elderly; musical training; neuroimagery and brain plasticity; psychometrics; executive function; mental health; well-being; sensorimotor function
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Longitudinal RCT (clinical trial) with an experimental group and an active control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- musical practice (Experimental): Intensive weekly musical keyboard training over 12 months
  Interventions: Behavioral: musical practice
- music education (Active Comparator): Recreative weekly musical courses without practice over 12 months
  Interventions: Behavioral: music education

INTERVENTIONS:
Behavioral: musical practice — Intensive weekly musical keyboard training over 12 months
  Arms: musical practice
Behavioral: music education — Recreative weekly musical courses without practice over 12 months
  Arms: music education

SUMMARY:
This longitudinal study aims to countervail age-related cognitive and cerebral decline in healthy retired people through intensive piano / keyboard music practice in Switzerland and Germany.

DETAILED DESCRIPTION:
Recent data suggest that music making might prevent cognitive decline in the elderly. However, experimental evidence remains sparse and no information on the neurophysiological basis has been provided, although cognitive decline is a major impediment to healthy aging. This study combines for the first time protocolled music practice in elderly with cutting-edge neuroimaging. The investigators propose a multi-site Hannover-Geneva longitudinal randomized intervention study in altogether 100 retired healthy elderly (64-76) years, 70 Geneva, 100 Hannover), offering either piano instruction or instruction on musical culture for one year. Participants will be tested at 3 time points on cognitive, perceptual and motor abilities as well as via wide-ranging functional and structural neuroimaging data (Magnetic Resonance Imaging, MRI). The research team expects positive transfer effects from intensive piano training not only on subjective well-being, but also on executive functions, working memory, hearing in noise and relationships of these behavioral features with morphological and functional brain plasticity. This study may therefore for the first time be demonstrate, that music making can provoke important societal impacts by diminishing cognitive and perceptual-motor decline underpinned by functional and structural brain plasticity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed volunteers, between 64 and 76 years of age, native French speakers. No regular musical practice over the lifespan. Only retired individuals may participate.

Exclusion Criteria:

* Impaired/not-corrected auditory or visual accuracy, neurological diseases in the present or the past, cardiovascular diseases, excessive hypertension, obesity, diabetes mellitus, beginning dementia, mild cognitive impairment, clinical depression.

Ages: 64 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Continuous Echo-Planar Imaging (EPI) | 18 months (4 measurements over time)
  Resting state functional Magnetic Resonance Imaging (MRI), informs on functional connectivity
Magnetization-Prepared 2 Rapid Acquisition Gradient Echo (MP2RAGE) | 18 months (4 measurements over time)
  Magnetic Resonance Imaging measure, allows to image gray matter
functional Magnetic Resonance Imaging (fMRI) | 18 months (4 measurements over time)
  Functional Imaging of a tonal Working Memory task, allows to study involved networks
Magnetic Resonance Diffusion Tensor Imaging (MR-DTI) | 18 months (4 measurements over time)
  Diffusion weighted echo-planar gradient echo sequence, allows to image white matter and structural connectivity
Magnetic Resonance Arterial Spin Labeling (MR-ASL) | 18 months (4 measurements over time)
  Blood perfusion assessment
Behavioral Battery (cognitive function) | 18 months (4 measurements over time)
  Comprehensive cognitive testing, full battery will be provided on request; involves Basic cognition, Executive Function, Fluid Intelligence, Verbal Memory

SECONDARY OUTCOMES:
Behavioral Battery (sensorimotor function) | 18 months (4 measurements over time)
  Sensorimotor testing, full battery will be provided on request; involves manual dexterity and hearing tests

CONTACTS AND LOCATIONS:
Overall Officials: Eckart Altenmüller, PhD, Principal Investigator — Hochschule für Musik, Theater und Medien Hannover
Locations (1):
- School of Health Sciences Geneva; HES-SO University of Applied Sciences and Arts Western Switzerland, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Raw (NIfTI format for MRI data) and preprocessed data will be made available to the scientific community, via an open source scientific data base.
Supporting Information: Study Protocol, SAP
Time Frame: December 2022
Access Criteria: Scientific community only

REFERENCES:
- [Derived] Losch H, Altenmuller E, Marie D, Passarotto E, Kretschmer CR, Scholz DS, Kliegel M, Kruger THC, Sinke C, Junemann K, James CE, Worschech F. Acquisition of musical skills and abilities in older adults-results of 12 months of music training. BMC Geriatr. 2024 Dec 19;24(1):1018. doi: 10.1186/s12877-024-05600-2. PMID 39702118
- [Derived] Mack M, Marie D, Worschech F, Kruger THC, Sinke C, Altenmuller E, James CE, Kliegel M. Effects of a 1-year piano intervention on cognitive flexibility in older adults. Psychol Aging. 2025 Mar;40(2):218-235. doi: 10.1037/pag0000871. Epub 2024 Dec 16. PMID 39679985
- [Derived] James CE, Altenmuller E, Kliegel M, Kruger THC, Van De Ville D, Worschech F, Abdili L, Scholz DS, Junemann K, Hering A, Grouiller F, Sinke C, Marie D. Train the brain with music (TBM): brain plasticity and cognitive benefits induced by musical training in elderly people in Germany and Switzerland, a study protocol for an RCT comparing musical instrumental practice to sensitization to music. BMC Geriatr. 2020 Oct 21;20(1):418. doi: 10.1186/s12877-020-01761-y. PMID 33087078